CLINICAL TRIAL: NCT05406193
Title: A New Care Model for Patients With Complicated Multimorbidity A Cluster-randomised Pilot Study in General Practice, Municipalities, and Hospitals
Brief Title: A New Care Model for Patients With Complicated Multimorbidity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Slagelse Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MM14
Record Dates: First submitted 2022-05-24; First posted 2022-06-06 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Multimorbidity
Keywords: General practice; Integrated care; Multimorbidity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (CIM2) (Experimental): An extended overview consultation, lasting 45 minutes, with the general practitioner, the patient (and maybe a relative), and the care coordinator. An individual care plan is developed, covering planned activities in the three sectors (general practice, municipality, and hospital) that will take place within the 12-month intervention period. General practice coordinates the planned patient care between general practice, the municipality, and the hospital, and follow-up on the execution of planned healthcare activities. The individual care plan is shared electronically with the healthcare center in the municipality and with the outpatient clinics using the standard IT-communication tool provided by MedCom and a routinely used national standard in general practice, hospitals, and municipalities.
  Interventions: Other: Patient-centred complex intervention in complicated multimorbidity (CIM2)
- Usual care (No Intervention): Patients with a general practitioner allocated to the control group will receive usual care.

INTERVENTIONS:
Other: Patient-centred complex intervention in complicated multimorbidity (CIM2) — CIM2 is the second version of the Patient-centred complex intervention in complicated multimorbidity
  Arms: Intervention (CIM2)

SUMMARY:
Patients with complex multimorbidity experience a high treatment burden, fragmentation of care and poor clinical outcomes. General practice is the key organizational setting in terms of offering these patients integrated, longitudinal, and patient-centered care. Therefore, we propose a new general practice based model to improve overview, patient involvement and integration of care. The new care model consist of a teaching session on multimorbidity for the health care professionals, a prolonged overview consultation for patients with complex multimorbidity with the general practitioner, resulting in an individual care plan shared with the municipalities and secondary care, access to cross-sectoral video conferences with secondary care specialists and. Control practices provide health care as usual. We evaluate the care model in a cluster-randomized non-blinded, parallel-group trial in general practice. Fourteen general practices are allocated 1:1 to either intervention or control. We evaluate the effectiveness of the intervention with patient-reported questionnaire at baseline, 6-month follow-up, and 12-month follow-up. Primary outcome measure is the Patient Assessment of Chronic Illness Care (PACIC). Secondary outcome measure includes patient-reported quality of life and the treatment burden for the patients with multimorbidity. Furthermore, the project include a process evaluation of the complex intervention with the objective to assess how the intervention is delivered and to identify important facilitators and barriers for implementing the intervention. The new model is integrated into the existing health care system structures and has the potential for a sustainable improvement in care for patients with complex multimorbidity.

ELIGIBILITY:
Inclusion Criteria:

1. Has more than one of the 3 common chronic diseases (diabetes, chronic obstructive pulmonary, chronic heart conditions)
2. Has been hospitalised, or visited an outpatient clinic due to their chronic diseases during the previous year
3. Take at least five different prescription drugs assessed from the Shared Medicine Card recording in the general practice
4. The general practitioner or the nurse in the practice recognise the patient as a "demanding" patient with complicated multimorbidity that will benefit from an overview consultation.

Exclusion Criteria:

* Patients who cannot speak Danish,
* Patients who cannot give informed consent,
* Patients who have a life expectancy of less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Patient Assessment of Chronic Illness Care (PACIC) at 12 months | From baseline to 12-month follow-up
  PACIC is a 20-item patient report instrument that assesses patient's receipt of clinical services and actions. Each item was scored on a 5-point scale ranging from 1 (no or never) to 5 (yes or always). Respondents rate how often they experienced the content described in each item. The scale range from 1-5 and is scored by averaging of items completed within that scale, and the overall PACIC is scored by averaging scores across all 20 items. Higher scores indicate higher patient assessment delivery of high-quality care for patients with chronic diseases.

SECONDARY OUTCOMES:
Change from baseline Patient Assessment of Chronic Illness Care (PACIC) at 6 months | From baseline to 6-month follow-up
  PACIC is a 20-item patient report instrument that assesses patient's receipt of clinical services and actions. Each item was scored on a 5-point scale ranging from 1 (no or never) to 5 (yes or always). Respondents rate how often they experienced the content described in each item. The scale range from 1-5 and is scored by averaging of items completed within that scale, and the overall PACIC is scored by averaging scores across all 20 items. Higher scores indicate higher patient assessment delivery of high-quality care for patients with chronic diseases.
Change from baseline EuroQol-5 Domain (EQ-5D-5L) at 6 months | From baseline to 6-month follow-up
  The EQ-5D-5L assess the patients' health-related quality of life. It contains two main elements: a descriptive profile comprising five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and the EQ-5D visual analogue scale (EQ VAS). Each dimension in the EQ-5D-5L has five response levels: no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5). The EQ-VAS range from 0 (the worst imaginable health state) at the bottom to 100 (the best imaginable health state) on the top for respondents to rate their overall health.
Change from baseline EuroQol-5 Domain (EQ-5D-5L) at 12 months | From baseline to 12-month follow-up
  The EQ-5D-5L assess the patients' health-related quality of life. It contains two main elements: a descriptive profile comprising five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and the EQ-5D visual analogue scale (EQ VAS). Each dimension in the EQ-5D-5L has five response levels: no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5). The EQ-VAS range from 0 (the worst imaginable health state) at the bottom to 100 (the best imaginable health state) on the top for respondents to rate their overall health.
Change from baseline Multimorbidity Treatment Burden Questionnaire (MTBQ) at 6 months | From baseline to 6-month follow-up
  The Multimorbidity Treatment Burden Questionnaire (MTBQ) is a 10-item questionnaire designed to measure treatment burden (the effort of looking after one's health) in patients with multimorbidity in primary care. Each question is scored as follows: zero (not difficult/ does not apply), one (a little difficult), two (quite difficult), three (very difficult), four (extremely difficult). To calculate a global score, each participant's average score is calculated from the questions answered and multiplied by 25 to give a score from 0-100. Higher MTBQ score indicate higher treatment burden.
Change from baseline Multimorbidity Treatment Burden Questionnaire (MTBQ) at 12 months | From baseline to 12-month follow-up
  The Multimorbidity Treatment Burden Questionnaire (MTBQ) is a 10-item questionnaire designed to measure treatment burden (the effort of looking after one's health) in patients with multimorbidity in primary care. Each question is scored as follows: zero (not difficult/ does not apply), one (a little difficult), two (quite difficult), three (very difficult), four (extremely difficult). To calculate a global score, each participant's average score is calculated from the questions answered and multiplied by 25 to give a score from 0-100. Higher MTBQ score indicate higher treatment burden.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Frølich, Professor, Study Chair — Innovation and Research Centre for Multimorbidity, Slagelse hospital, Region Zealand
Locations (11):
- Denmark (11):
  - Lægerne Kanaltorvet, Albertslund
  - Thorkil Christensen, Albertslund
  - Brøndbyøster Torv, Brøndby
  - Lægerne i Brohuset, Ishøj
  - Lægecenter Korsør, Korsør
  - Læge Depenau vej-Hansen, Slagelse
  - Læge Jørgen Larsen, Slagelse
  - Læge Lene Stiggaard, Slagelse
  - Lægerne Reventlow, Wolfhagen og Bendtsen, Slagelse
  - Lægerne ved Lystskoven, Slagelse
  - Lægerne Vallensbæk Nord, Vallensbæk

REFERENCES:
- [Derived] Lundstrom SL, Kamstrup-Larsen N, Barrett BA, Jorgensen LMB, Hansen SS, Andersen JS, Friderichsen B, Stockmarr A, Frolich A. A patient-centred care model for patients with complicated multimorbidity: Protocol for a pilot cluster randomised trial in general practice, municipalities, and hospitals. PLoS One. 2024 Dec 4;19(12):e0310697. doi: 10.1371/journal.pone.0310697. eCollection 2024. PMID 39630823

DOCUMENTS (1):
  • Study Protocol (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/93/NCT05406193/Prot_000.pdf